## DynaSSaur

## **Consent form: People with CF**

| Full study name: | | Dynamic Chest X-ray with Simultaneous Spirometry | |
|---|---|---|---|
| IRAS: | | 322890 | |
| Principal investigator:<br>Co-investigators: | | Dr David Green<br>Professor Martin Walshaw<br>Dr Dilip Nazareth<br>Dr Freddy Frost | |
| | | | Please<br>initial box |
| 1. | . I confirm that I have read the Participant Information Sheet dated 20/09/2023 (version 3.1) for the above study. I have had the opportunity to consider the information, ask questions, and have had these answered satisfactorily. | | |
| 2. | 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, and without my medical care or legal rights being affected. | | |
| 3. | I understand that my data will be stored securely on NHS servers or within locked areas of LHCH, in line with NHS data protection regulations, GDPR (General Data Protection Regulation), and DPA (Data Protection Act 2018). GDPR and The DPA are designed to regulate how data should be handled appropriately to protect personalised information. | | |
| 4. | | draw from this study, the researchers may keep my information for nely keep this information for up to 20 years. | |

Version 3.1 Date 20/09/2023

Page **1** of **2** 

| Nan | ne of participant | Date | Signature | |
|---|---|---|---|---|
| 9. | <ol> <li>I understand that any information I write in the questionnaire 'free text' box may be published,<br/>in a completely anonymous form, by the study team.</li> </ol> | | | |
| 8. | 8. I agree to take part in the above study, which will involve a review of my medical notes a well as attending LHCH for a dynamic chest X-ray and spirometry (breathing tests). | | • | ; |
| 7. | me or provide information a | bout my health status. As | d by LHCH may be used to help contact part of this, I understand that my GP hey need to know or act upon. | |
| 6. | I understand that the inform the future and may be share | | will be used to support other research in er researchers. | |
| | | ers of the study team whe | ere it is relevant to my taking part in this | |
| 5. | Lunderstand that relevant so | ections of my medical no | es and data collected during the study | |

One copy of this consent form is to be stored securely in the Site Investigator File.

One copy of this consent form is to be provided to the participant.

Version 3.1 Date 20/09/2023